CLINICAL TRIAL: NCT03515200
Title: A Phase I Study of Palbociclib in Combination With Chemotherapy in Pediatric Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia
Brief Title: Treatment With Combination Chemotherapy for Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to departure of PI from St. Jude
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RELPALL; NCI-2018-00814 (Registry Identifier: [Registry ID: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2018-04-19; First posted 2018-05-03 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphoblastic Leukemia With Failed Remission
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — palbociclib; Methotrexate; Dexamethasone; Calcium Dobesilate; Bortezomib; Dasatinib; Doxorubicin; ruxolitinib

STUDY DESIGN:
Intervention Model Description: Palbociclib will be administered orally on Days 1-5, and 11-15 concurrently with dexamethasone of each 30 day cycle for one cycle (dose escalation) or up to 3 cycles for responders (dose expansion). Bortezomib will be given on Days 7, 10, 17 and 20. Doxorubicin will be given on Days 7 and 17. If the dose escalation with this schema is tolerated, a final dose level administering additional doses of palbociclib on days 21-30 will be evaluated.
  Patients with Ph-like or Ph+ ALL will receive tyrosine kinase inhibitor (TKI) beginning on Day 7.
  Triple intrathecal chemotherapy (MHA) will be given on Day 1 of the course. The frequency and total number of IT MHA is based on the patient's level of CNS disease.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): This study will be done in two parts: Part 1: Dose escalation and Part 2: Dose expansion.
  In Part 1 - Dose escalation: Patients that lack Ph+ or Ph-like ALL, palbociclib, initially at 50mg/m2/day, 40% of the adult MTD, will be administered on Days 1-5 and 11-15, and escalated based on tolerability. If our highest dosing of 100mg/m2/day is tolerated, we will have a final dose level that receives an additional 10 days of palbociclib (Days 1-5, 11-15, and 21-30).
  For patients that are Ph+ or have Ph-like ALL that are also receiving dasatinib or ruxolitinib: palbociclib, initially at 75mg/m2/day, 60% of the adult MTD, will be administered on Days 1-5 and 11-15 and escalated based on tolerability.
  In Part 2 - Dose expansion: After determination of dose in Part 1, an additional 10 patients will be enrolled to confirm tolerability.
  Interventions: Drug: Palbociclib Oral Capsule; Drug: Intrathecal Triple Therapy; Drug: Dexamethasone; Drug: Bortezomib; Drug: Dasatinib; Drug: Doxorubicin; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Palbociclib Oral Capsule — Given orally or nasogastrically (NG).
  Other Names: Ibrance®
Drug: Intrathecal Triple Therapy — Given intrathecally (IT).
  Other Names: ITMHA; methotrexate/hydrocortisone/cytarabine
Drug: Dexamethasone — Given orally, nasogastrically (NG) or intravenously (IV).
  Other Names: Decadron
Drug: Bortezomib — Given intravenously (IV) or subcutaneously (SC).
  Other Names: Velcade®
Drug: Dasatinib — Given orally or nasogastrically (NG).
  Other Names: Sprycel®
Drug: Doxorubicin — Given intravenously (IV).
  Other Names: Adriamycin®
Drug: Ruxolitinib — Given orally or nasogastrically (NG).
  Other Names: Jakafi®

SUMMARY:
Leukemia cells grow and divide fast and out of control. In normal cells, certain proteins called CDK4 and CDK6 control cell growth. The study drug called palbociclib works by blocking the CDK4 and CDK6 proteins. Palbociclib has been shown to kill leukemia cells in the laboratory and in animal studies. Palbociclib will be added to other chemotherapy drugs, such as dexamethasone, that are known to be effective in treating childhood ALL.

This study will be done in two parts: Part 1: Dose Escalation and Part 2: Dose Expansion. The goal of Part 1 of the study is to find the highest tolerable combination of palbociclib and chemotherapy that the investigators can give to patients with leukemia. Once those doses are determined, the investigators will enroll patients on Part 2: Dose Expansion. This phase will enroll additional patients that receive the highest tolerated dose of palbociclib as determined in part 1, in order to better understand the side effects and how effective this treatment approach is.

With this research study, the investigators hope to meet the following goals:

* To find the highest tolerable dose of palbociclib in combination with chemotherapy that can be given without causing severe side effects;
* To learn what kind of side effects palbociclib in combination with chemotherapy may have; and
* To learn more about the biology effects of palbociclib on the cells in the participant's body.

Up to 40 children, adolescents and young adults will participate in both parts of this study at St. Jude only.

DETAILED DESCRIPTION:
RELPALL is a single center, St Jude initiated, non-randomized single-arm phase I study to characterize the toxicity profile and to determine the maximum tolerated combination (MTC) and recommended phase II combination of palbociclib when given with chemotherapy in pediatric patients with relapsed or refractory acute lymphoblastic leukemia (ALL). Palbociclib is a reversible inhibitor of cyclin-dependent kinase 4 (CDK4) and the closely related cyclin-depending kinase 6 (CDK6) that has shown high anti-leukemic activity in several pre-clinical models. The mechanism of palbociclib, which reversibly arrests cells in G1, argues that combination treatment, as opposed to single agent treatment, will be more likely to provide clinical benefit. Timing of combination treatment with standard cytotoxic chemotherapy drugs that kill actively dividing cells is important to maximize the chance of activity. This study will build on prior multiple myeloma experience with palbociclib in combination with dexamethasone and bortezomib while tailoring the treatment to pediatric relapsed/refractory ALL. To maximize G1 arrest, dexamethasone will be given concurrently with palbociclib for five days. Patients will receive a 48 hour "washout" before receiving bortezomib and doxorubicin, both cytotoxic anti-leukemic drugs that preferentially kills cells when synchronized in S phase. Patients with Philadelphia Chromosome positive ALL (Ph+) and Philadelphia-like (Ph-like) ALL will also receive a tyrosine kinase inhibitor (TKI) beginning on Day 7 until count recovery. The primary objective is to determine a tolerable combination of palbociclib plus chemotherapy in pediatric patients with relapsed or refractory ALL. The secondary objective is to estimate the overall response rate to the combination of palbociclib and chemotherapy in pediatric patients with relapsed or refractory ALL. Exploratory objectives include measuring cell cycle kinetics of ALL cells following administration of palbociclib and an evaluation of modes of resistance in non-responders.

ELIGIBILITY:
Inclusion Criteria:

Participants must be < 22 years of age.

Diagnosis:

Participants must have a diagnosis of acute lymphoblastic leukemia and disease meets at least one of the following criteria:

* relapsed or refractory to chemotherapy as defined by ≥5% leukemic blasts in the bone marrow or flow cytometry confirmed leukemic blasts in the peripheral blood
* relapsed after hematopoietic stem cell transplantation (HSCT)

Patients must have had histologic, morphologic or flow cytometric verification of the malignancy at relapse.

Performance Level:

Karnofsky or Lansky performance score is ≥ 50% (corresponding to ECOG Score of ≤ 2). The Lansky performance score should be used for participants < 16 years and the Karnofsky performance score for participants ≥ 16 years. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

Prior Therapy:

Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study.

Patients who relapse on therapy other than standard ALL maintenance must have fully recovered from the acute toxic effects of all prior anti-cancer therapy, defined as resolution of all such toxicities to ≤ Grade 2 or lower per the inclusion/exclusion criteria prior to entering this study.

At least 14 days must have elapsed since the completion of cytotoxic therapy, with the exception of standard maintenance therapy and steroids.

At least 7 days must have elapsed since completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period prior to enrollment must be extended beyond the time during which adverse events are known to occur.

At least 3 half-lives must have elapsed since prior therapy that included a monoclonal antibody with the exception of blinatumomab. Patients must have been off blinatumomab infusion for at least 7 days and all drug related toxicity must have resolved to grade 2 or lower as outlined in the inclusion/exclusion criteria.

At least 42 days must have elapsed since CAR-T cell therapy.

At least 90 days have elapsed since bone marrow transplant and participant is off immune suppression for ≥ 2 weeks, if applicable with no evidence of active GVHD.

At least 2 weeks must have elapsed since local XRT (small port); ≥ 3 months must have elapsed if prior cranial or craniospinal XRT was received, if ≥ 50% of the pelvis was irradiated, or if TBI was received; ≥ 6 weeks must have elapsed if other substantial bone marrow irradiation was given.

Organ Function Requirements:

Adequate renal function defined as glomerular filtration rate ≥ 60 cc/min/1.73m2 or serum creatinine based on age as follows:

* Age: <6 months; maximum serum creatinine (mg/dL): 0.4 (male, female); Age: 6 months to <1 year; maximum serum creatinine (mg/dL): 0.5 (male, female); Age: 1 to < 2 years; maximum serum creatinine (mg/dL): 0.6 (male, female); Age: 2 to < 6 years; maximum serum creatinine (mg/dL): 0.8 (male, female); Age: 6 to <10 years; maximum serum creatinine (mg/dL): 1 (male, female); Age: 10 to <13 years; maximum serum creatinine (mg/dL): 1.2 (male, female); Age: 13 to <16 years; maximum serum creatinine (mg/dL): 1.5 (male), 1.4 (female); Age: ≥ 16 years; maximum serum creatinine (mg/dL): 1.7 (male), 1.4 (female)

Adequate hepatic function defined as:

* Total bilirubin ≤ 2 x upper limit of normal (ULN) for age, and
* ALT ≤ 3 x ULN for age, unless elevation is due to leukemic infiltration.

Adequate cardiac function defined as shortening fraction of ≥ 27% or ejection fraction ≥ 45%.

Adequate pulmonary function defined as:

* No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94%.
* No evidence of acute pulmonary infiltrates on chest radiograph.

Adequate central nervous system (CNS) function defined as:

* Patients with seizure disorder may be enrolled if on allowed anti-convulsants and well controlled. Benzodiazepines and gabapentin are acceptable.
* CNS toxicity < Grade 2

Adequate peripheral nervous system (PNS) function defined as:

* PNS toxicity < Grade 2.

Exclusion Criteria:

Extramedullary disease status: patients with isolated CNS disease or isolated testicular disease are not eligible.

Concurrent chemotherapy or targeted anti-cancer agents, other than intrathecal therapy.

Patients who have previously received bortezomib or other proteasome inhibitors that did not have a response while receiving the inhibitor are not eligible. Patients that responded but had a subsequent relapse are eligible.

Patients who have previously received palbociclib or other CDK4/6 inhibitors are not eligible.

Patient with concurrent severe and/or uncontrolled medical conditions that, in the opinion of the investigator, may impair participation in the study or the evaluation of safety and/or efficacy.

Patients that have an active, uncontrolled infection are not eligible.

Known HIV infection or active hepatitis B (defined as hepatitis B surface antigen-positive) or C (defined as hepatitis C antibody-positive).

Pregnant or lactating (female participant of childbearing potential must have negative serum or urine pregnancy test required within 7 days prior to start of treatment).

Male or female participant of reproductive potential must agree to use appropriate methods of contraception for the duration of study treatment and for at least 30 days after last dose of protocol treatment.

Cumulative anthracyclines must not exceed 450mg/m2 doxorubicin equivalents following completion of treatment on protocol. Therefore for patients receiving one course on protocol cumulative anthracyclines must be less than or equal to 400mg/m2 doxorubicin equivalents at the time of enrollment

Inability or unwillingness or research participant or legal guardian/representative to give written informed consent.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2018-04-20 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of palbociclib plus chemotherapy | End of cycle 1 (day 40 of therapy)
  Determine a tolerable combination of palbociclib plus chemotherapy in pediatric patients with relapsed or refractory ALL.

SECONDARY OUTCOMES:
Treatment response | During the dose expansion phase, following completion of chemotherapy doses and prior to the subsequent course up to 3 cycles, if applicable (each cycle is 30 days)
  percentage of patients who attain complete remission (CR)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja A. Gruber, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols